CLINICAL TRIAL: NCT07219251
Title: Engagement of Veterans With Lung Cancer (EVLC)
Brief Title: Engagement of Veterans With Lung Cancer
Acronym: EVLC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto Veterans Institute for Research (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Manali Patel, Staff Oncologist and Investigator, VA Palo Alto Health Care System
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: IRB-79923; LC240650 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2025-10-02; First posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Lung Cancer (NSCLC); Lung Adenocarcinoma; Lung Cancer, Non-Small Cell; Lung Carcinoma; Lung Cancer, Small Cell; Lung Adenocarcinoma With Bronchiolo-alveolar Feature
Keywords: lung; cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Small Cell Lung Carcinoma; Neoplasms

STUDY DESIGN:
Intervention Model Description: intervention vs. usual care
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The statistician analyzing the data will be masked from the randomization assignment. The principal investigator overseeing the trial will have access to the data but will also be masked from randomization assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care - Arm A (Active Comparator): Patients randomized to this group will receive usual care provided by their oncology(or primary) clinical team.
  Interventions: Other: Usual Care Group
- Intervention Lay Health Worker (LHW) - Arm B (Experimental): Participants randomized to this arm of the study will receive usual care with supplemental education and support provided by a lay health worker (LHW) to assist with healthcare planning, symptom management, and discussions about care preferences and goals.
  Interventions: Behavioral: Lay Health Worker (LHW) Planning

INTERVENTIONS:
Behavioral: Lay Health Worker (LHW) Planning — Patients randomized to the LHW group will receive usual care provided by their oncology (or primary) clinical team along with an initial 30-minute telephone call with the LHW from Palo Alto, followed by weekly 15-minute phone calls (or as needed) for 6months. These calls are designed to assist with healthcare planning, symptom management, and discussions about care preferences and goals.
  Arms: Intervention Lay Health Worker (LHW) - Arm B
Other: Usual Care Group — Participants randomized to the usual care group will receive usual care provided by their oncology clinical team. These teams have been trained in symptom assessment, goals-of-care (GoC) discussions, and documentation of such clinical services. As part of usual care, participants may engage in symptom and GoC discussions at any time, initiated by either the patient or the clinician.
  Other Names: Usual Care
  Arms: Usual Care - Arm A

SUMMARY:
This research study will help our understanding of whether additional support for Veterans with lung cancer can improve their quality of life.

DETAILED DESCRIPTION:
This study aims to evaluate whether a lay health worker who provides education and support regarding goals of care and symptom management can improve health-related quality of life among Veterans with newly diagnosed lung cancer and those receiving treatment or who have completed treatment within 12 months as compared to usual care. We will also determine whether the intervention reduces acute care use and explore effects on anxiety and depression, patient activation, and goals of care communication. This knowledge is important as it will help to improve care for Veterans with lung cancer.

PRIMARY OBJECTIVES:

i.) Health-related quality of life

SECONDARY OBJECTIVES:

i.) acute care use ii.) patient activation iii.) anxiety and depression iv.) documentation of goals of care (GoC) v.) palliative care use vi.) hospice use

OUTLINE: The study will enroll and randomize 1:1 a total of 194 Veterans diagnosed with lung cancer (any stage).

Arm A: Participants randomized to the usual care group will receive usual care provided by their oncology clinical team.

Arm B: Participants randomized to the LHW group will receive usual care provided by their oncology clinical team and also receive weekly telephone calls with a trained lay health worker to assist with healthcare planning, symptom management, and discussions about care preferences and goals for 6 months.

All participants regardless of group randomization, will be required to complete surveys at the start of the study and at 3-month intervals for 12 months (i.e., at enrollment, 3 months, 6 months, 9 months, and 12 months).

ELIGIBILITY:
Inclusion Criteria:

1. Veteran patients with diagnosis of any stage of lung cancer;
2. 18 years of age or older;
3. English- or Spanish-speaking;
4. can self-administer questionnaires in English or Spanish;
5. valid telephone number;
6. receiving oncology care at participating sites;
7. currently newly diagnosed or receiving or having completed systemic anti-cancer therapy and/or radiation therapy within 12 months, defined as oral, injection, or intravenous therapy (chemotherapy, targeted therapy, or immunotherapy)

Exclusion Criteria:

1. no capacity to consent;
2. actively receiving hospice care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2025-10-25 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Health-Related Quality of Life | At Baseline (time of enrollment), 3, 6, 9, and 12 months post-enrollment
  Change in Health-related quality of life using the 36-item validated Functional Assessment of Cancer Therapeutics-Lung (FACT-L) survey.

SECONDARY OUTCOMES:
Emergency Department Visits (Self-reported and Chart Review) | From baseline (time of enrollment) to 12 Months post-enrollment
  Emergency Department use will be self-reported by each patient or abstracted by electronic medical record at 3, 6, 9 and 12 months after enrollment.
Hospitalization Visits (Self-reported and Chart Review) | From baseline (time of enrollment) to 12 months post-enrollment
  Hospital use for each patient will be self-reported by each patient or abstracted by electronic medical record at 3, 6, 9 and 12 months after enrollment.
Patient Activation Measure (PAM-10). | At baseline (time of enrollment), 3, 6, 9 and 12 months post-enrollment
  Change in patient activation using 10-item validated survey Patient Activation Measure (PAM-10) assessing patient activation in their health and health care .
Patient-reported anxiety and depression | At baseline, 3, 6, 9 and 12 months post-enrollment
  Patient-reported anxiety and depression using the validated Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety and Depression scales
Documentation of goals of care discussions (Chart Review) | At baseline, 3, 6, 9 and 12 months post-enrollment
  Documentation of goals of care discussions will be abstracted by electronic medical record chart review for each patient at 3, 6, 9 and 12 months after enrollment.
Palliative Care Use (Self-reported and Chart Review) | From baseline (time of enrollment) to 12 months post-enrollment
  Palliative care use will be self-reported by each patient or abstracted by electronic medical record at 3, 6, 9 and 12 months after patient enrollment.
Hospice Care Use (Self-reported and Chart Review) | From baseline (time of enrollment) to 12 months post-enrollment
  Hospice care use will be self-reported by each patient or abstracted by electronic medical record at 3, 6, 9 and 12 months after patient enrollment.

CONTACTS AND LOCATIONS:
Locations (1):
- Veterans Affairs Palo Alto Health Care System (VAPAHCS), Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No